CLINICAL TRIAL: NCT03424707
Title: A Single-Center, Randomized, Double-Blind, Parallel, Pilot Study to Evaluate the Efficacy and Safety of Fixed Dose Combination of DW340 in Patients With Acute Low Back Pain
Brief Title: A Study to Evaluate the Efficacy and Safety of Fixed Dose Combination of DW340 in Patients With Acute Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DW340-P2
Record Dates: First submitted 2018-01-31; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Acute Low Back Pain
MeSH Terms: interventions — eperisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combination (Experimental)
  Interventions: Drug: DW340(pelubiprofen/eperisone)
- single (Active Comparator)
  Interventions: Drug: Pelubi(pelubiprofen)
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: DW340(pelubiprofen/eperisone) — DW340
  Arms: combination
Drug: Pelubi(pelubiprofen) — pelubiprofen
  Arms: single
Drug: Placebo Oral Tablet — Placebo Oral Tablet
  Arms: placebo

SUMMARY:
A Single-Center, Randomized, Double-Blind, Parallel, Pilot Study to Evaluate the Efficacy and Safety of Fixed Dose Combination of Pelubiprofen/Eperisone in Patients with Acute Low Back Pain

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years of age
2. Patients with a paraxial (muscle spasm) of less than 21 days and acute lower back pain. Randomized intervention. Arterial pain 100 mm - visual analogue scale (VAS)
3. Participation and voluntary agreement

Exclusion Criteria:

1. Drugs for Clinical Trial or Similar Drugs and Components with Hypersensitivity or Aspirin or Nonsteroidal Anti-inflammatory Drugs
2. Those accompanying the following diseases (1) patients with severe underlying diseases that cause back pain (eg, cancer, spinal infections, cauda equina syndrome, spinal stenosis, neuropathy, vertebral compression fracture, posterior hiatal joint syndrome, intervertebral disc herniation, fibromyalgia, Spondylolisthesis, imaging confirmed degenerative spondylosis, severe arthritis or severe osteoporosis) (2) myositis, muscular atrophy, myotonia, myasthenia (3) peptic ulcer or duodenal ulcer (4) Gastrointestinal bleeding or bleeding disorder (5) severe heart failure (NYHA class III / IV) (6) Uncontrolled hypertension (SBP ≥ 180 mmHg or DBP ≥ 110 mmHg) (7) Liver impairment (AST or ALT ≥ 3 × upper normal level of the organ) or renal impairment (CLcr <30 mL / min)
3. Those who have confirmed the following history or surgery / (1) lumbar surgery (2) Unstable angina pectoris, myocardial infarction, transient ischemic attack, stroke, coronary artery bypass surgery or coronary artery bypass graft within 6 months from screening (3) galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption, (4) malignant tumor within 5 years from the screening point
4. Drugs that may affect the following efficacy evaluations during clinical trials, or those expected to require drug interactions with the clinical trial drug (provided there is a separate standard, such as a nonsteroidal anti-inflammatory drug) Follow the standard.) (1) Nonsteroidal antiinflammatory drugs: pelubiprofen, aceclofenac, diclofenac, ketorolac (from 1 week before randomization until the end of the clinical trial, except oxaprozin and oxicam 2 weeks before randomization) (2) Muscle relaxants: eperisone, baclofen, cyclobenzaprine, dantrolene, thiocolchicoside, tizanidine (from 1 week before randomization until the end of the study) (3) Analgesics: acetaminophen (paracetamol), codeine, oxycodone, tramadol, etc. (However, in the case of narcotic analgesics, (4) systemic or low back pain or steroids (from 4 weeks prior to randomization until the end of the study) (5) Contraindications during other clinical trials Drug / taboo treatment (see 7.4)
5. Pregnant or lactating women and appropriate contraceptive *

   * Use of hormonal contraceptive, intrauterine devices, spouse sterilization (vasectomy, tubal ligation, etc.), double blockage (use of spermicide in combination with vaginal septum, vaginal sponge or neck cap)
6. Those who have received other clinical trial drugs within a longer period of 12 weeks or more than half of the half-life before screening
7. Those who are unable to participate in the clinical trial according to the testee's judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
100mm VAS | 7 days
  The change of 100mm movement pain VAS between basline and end point